CLINICAL TRIAL: NCT01325051
Title: A Phase IV, Open-Label Study to Characterize the First-Dose and Multiple-Dose Pharmacokinetics of Raltegravir in the Gastrointestinal Tract of Healthy Male Volunteers
Brief Title: Study to Characterize the Pharmacokinetics of Raltegravir in the Gastrointestinal (GI) Tract of Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Angela Kashuba, PharmD (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor-Investigator, Angela Kashuba, PharmD, Associate Professor, University of North Carolina, Chapel Hill
Organization: University of North Carolina, Chapel Hill (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CID 1020; IRB 10-2321
Record Dates: First submitted 2011-03-23; First posted 2011-03-29 (Estimated); Last update posted 2012-01-05 (Estimated); Status verified 2012-01

CONDITIONS: Healthy Volunteer
Keywords: raltegravir; pharmacokinetics; healthy; male; volunteers; gastrointestinal; tract
MeSH Terms: interventions — Raltegravir Potassium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Raltegravir (No Intervention): To test raltegravir to see if it can be detected in gastrointestinal tissue of healthy men.
  Interventions: Drug: Raltegravir

INTERVENTIONS:
Drug: Raltegravir — 400 mg tablets by mouth BID from Day 1 - Day 7 after enrollment visit
  Other Names: MK-0518; ISENTRESS

SUMMARY:
The purpose of this study is to characterize the way the first commercially available integrase inhibitor, raltegravir, a new class of antiretrovirals that is used to treat HIV, is distributed into the rectal mucosal tissue. This information will generate important information regarding the drug's penetration into lymphoid tissues that are rapidly depleted in HIV infection. Subsequently strategies to prevent the sexual transmission of HIV and for treating HIV-infected individuals will be designed.

DETAILED DESCRIPTION:
Participants: 14 HIV-uninfected, healthy, male volunteers, ≥18 and ≤49 years of age, will be recruited and enrolled. Healthy is defined as no clinically relevant abnormalities identified by a detailed medical history, full physical examination, including blood pressure and pulse rate measurement, 12-lead ECG, and clinical laboratory tests. Participants of all races and ethnicities will be considered for enrollment. This study will be conducted at a single site in the United States: the University of North Carolina at Chapel Hill.

Procedures (methods): An outpatient screening visit will be conducted on all potential participants to obtain informed consent and evaluate for eligibility. Once enrolled, all subjects will take 400 mg oral dose of raltegravir twice daily from Day 1 to Day 7. The healthy men enrolled in this study will undergo single-dose and multiple-dose pharmacokinetic sampling. Blood will be collected via peripheral IV at pre-dose, and at 1, 2, 3, 4, 6, 8 and 12 hours post-dose. Subjects will undergo two colonoscopies during sampling visits (Day 1 and Day 7) for the purpose of obtaining gastrointestinal-associated lymphoid tissue (GALT). Each subject will have his biopsy obtained at one of the following time points post-dose: 1, 2, 3, 4, 6, 8, and 12 hours. Seven to ten days after their last inpatient sampling visit, all subjects will complete a follow-up visit.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male subjects between the ages of 18 and 49 years, inclusive, with intact genital tract and gastrointestinal tract. Healthy is defined as no clinically relevant abnormalities identified by a detailed medical history, full physical examination, including blood pressure and pulse rate measurement, 12-lead ECG, and clinical laboratory tests.
2. Body Mass Index (BMI) of approximately 18 to 30 kg/m^2; and a total body weight greater than or equal to 50 kg (110 lbs).
3. Evidence of a personally signed and dated informed consent document indicating that the subject has been informed of all pertinent aspects of the trial.
4. Willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other trial procedures.

Exclusion Criteria

1) any medical condition or finding deemed by the investigators to be ineligible

Ages: 18 Years to 49 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2011-04; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
AUC = Area under the concentration versus time curve of raltegravir | 0, 1, 2, 3, 4, 6, 8, and 12 hours after single dose (Day 1) and 0, 1, 2, 3, 4, 6, 8, and 12 hours after 13 doses (Day 7)

SECONDARY OUTCOMES:
Cmax = maximum concentration of raltegravir | 0, 1, 2, 3, 4, 6, 8, and 12 hours after single dose (Day 1) and 0, 1, 2, 3, 4, 6, 8, and 12 hours after 13 doses (Day 7)
Tmax = time to maximum concentration of raltegravir | 0, 1, 2, 3, 4, 6, 8, and 12 hours after single dose (Day 1) and 0, 1, 2, 3, 4, 6, 8, and 12 hours after 13 doses (Day 7)
C12 = concentration at 12 hours after dose of raltegravir | 0, 1, 2, 3, 4, 6, 8, and 12 hours after single dose (Day 1) and 0, 1, 2, 3, 4, 6, 8, and 12 hours after 13 doses (Day 7)
t1/2 = half-life of raltegravir | 0, 1, 2, 3, 4, 6, 8, and 12 hours after single dose (Day 1) and 0, 1, 2, 3, 4, 6, 8, and 12 hours after 13 doses (Day 7)

CONTACTS AND LOCATIONS:
Overall Officials: Angela Kashuba, PharmD, Principal Investigator — UNC-CH School of Pharmacy; Kristine Patterson, MD, Principal Investigator — UNC-CH Division of Infectious Diseases
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

REFERENCES:
- [Background] Musicco M, Lazzarin A, Nicolosi A, Gasparini M, Costigliola P, Arici C, Saracco A. Antiretroviral treatment of men infected with human immunodeficiency virus type 1 reduces the incidence of heterosexual transmission. Italian Study Group on HIV Heterosexual Transmission. Arch Intern Med. 1994 Sep 12;154(17):1971-6. PMID 8074601
- [Background] Otten RA, Smith DK, Adams DR, Pullium JK, Jackson E, Kim CN, Jaffe H, Janssen R, Butera S, Folks TM. Efficacy of postexposure prophylaxis after intravaginal exposure of pig-tailed macaques to a human-derived retrovirus (human immunodeficiency virus type 2). J Virol. 2000 Oct;74(20):9771-5. doi: 10.1128/jvi.74.20.9771-9775.2000. PMID 11000253
- [Background] Lallemant M, Jourdain G, Le Coeur S, Mary JY, Ngo-Giang-Huong N, Koetsawang S, Kanshana S, McIntosh K, Thaineua V; Perinatal HIV Prevention Trial (Thailand) Investigators. Single-dose perinatal nevirapine plus standard zidovudine to prevent mother-to-child transmission of HIV-1 in Thailand. N Engl J Med. 2004 Jul 15;351(3):217-28. doi: 10.1056/NEJMoa033500. Epub 2004 Jul 9. PMID 15247338
- [Background] Blankson JN, Persaud D, Siliciano RF. The challenge of viral reservoirs in HIV-1 infection. Annu Rev Med. 2002;53:557-93. doi: 10.1146/annurev.med.53.082901.104024. PMID 11818490
- [Background] Pierson T, Hoffman TL, Blankson J, Finzi D, Chadwick K, Margolick JB, Buck C, Siliciano JD, Doms RW, Siliciano RF. Characterization of chemokine receptor utilization of viruses in the latent reservoir for human immunodeficiency virus type 1. J Virol. 2000 Sep;74(17):7824-33. doi: 10.1128/jvi.74.17.7824-7833.2000. PMID 10933689
- [Background] Isentress (raltegravir) Prescribing Guide. Merck & Co, Inc. October 2007.
- [Background] Markowitz M, Morales-Ramirez JO, Nguyen BY, Kovacs CM, Steigbigel RT, Cooper DA, Liporace R, Schwartz R, Isaacs R, Gilde LR, Wenning L, Zhao J, Teppler H. Antiretroviral activity, pharmacokinetics, and tolerability of MK-0518, a novel inhibitor of HIV-1 integrase, dosed as monotherapy for 10 days in treatment-naive HIV-1-infected individuals. J Acquir Immune Defic Syndr. 2006 Dec 15;43(5):509-15. doi: 10.1097/QAI.0b013e31802b4956. PMID 17133211
- [Background] Barau C, Delaugerre C, Braun J, de Castro N, Furlan V, Charreau I, Gerard L, Lascoux-Combe C, Molina JM, Taburet AM. High concentration of raltegravir in semen of HIV-infected men: results from a substudy of the EASIER-ANRS 138 trial. Antimicrob Agents Chemother. 2010 Feb;54(2):937-9. doi: 10.1128/AAC.01261-09. Epub 2009 Dec 7. PMID 19995925